CLINICAL TRIAL: NCT00343291
Title: Phase II Randomized, Open-Label Study of Cetuximab and Bevacizumab in Combination With Paclitaxel and Carboplatin in Patients With Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: A Study of Cetuximab and Bevacizumab in Combination With Paclitaxel and Carboplatin in Stage IIIb/IV NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13421; I4E-MC-S001 (Other: Eli Lilly and Company); CP02-0554 (Other: ImClone)
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Malignant pleural effusions
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant | interventions — Cetuximab; Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) (Active Comparator): Cycles 1-6:
  * Cetuximab 400 mg/m² initial dose on day 1 and then 250 mg/m² given every week
  * Bevacizumab 15 mg/kg given on day 8 of every 3 week cycle
  * Paclitaxel 200 mg/m² on day 1 of every 3 week cycle
  * Carboplatin area under curve (AUC=6 min*mg/mL) on day 1 of every 3 week cycle
  Patients who demonstrate a response or stable disease after six cycles of therapy may continue on weekly cetuximab monotherapy until disease progression, unacceptable toxicity, or another withdrawal criterion is met
  Interventions: Biological: Cetuximab; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3) (Active Comparator): Cycles 1-6:
  * Cetuximab 400 mg/m² initial dose on day 1 and then 250 mg/m² given every week
  * Bevacizumab 15 mg/kg given on day 8 of every 3 week cycle
  Cycles 1-3:
  * Paclitaxel 200 mg/m² on day 1 of each 3 week cycle for the first 3 cycles
  * Carboplatin AUC=6 min*mg/mL on day 1 of each 3 week cycle for the first 3 cycles
  Patients who demonstrate a response or stable disease after six cycles of therapy may continue on weekly cetuximab monotherapy until disease progression, unacceptable toxicity, or another withdrawal criterion is met
  Interventions: Biological: Cetuximab; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Cetuximab — Administered intravenously
  Other Names: Erbitux
Biological: Bevacizumab — Administered intravenously
Drug: Paclitaxel — Administered intravenously
Drug: Carboplatin — Administered intravenously

SUMMARY:
The primary objective of this study will be to determine the progression free survival of patients with stage IIIb/IV non-small cell lung cancer (NSCLC) treated with dual agent monoclonal antibody therapy consisting of cetuximab and bevacizumab in combination with two different regimens of paclitaxel and carboplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient has histologically or cytologically confirmed non-small cell lung cancer (NSCLC), except squamous cell carcinoma. Mixed tumors will be categorized by the predominant cell type, but the presence of small cell lung cancer elements will make the patient ineligible. Cytologic or histologic elements can be established on metastatic tumor aspirates or biopsy.
* The patient has advanced NSCLC (Stage IIIB with malignant pleural effusion or Stage IV or recurrent disease).
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST).
* The patient's Eastern Cooperative Oncology Group (ECOG) performance status is 0 or 1.
* The patient has adequate hematologic function as defined by an Absolute Neutrophil Count greater than or equal to 1500/mm³,hemoglobin greater than or equal to 9 gm/dL, and a platelet count greater than or equal to 100,000/mm³ obtained within 2 weeks prior to the first dose of study medication.
* The patient has adequate hepatic function as defined by a total bilirubin greater than or equal to 1.5 mg/dL and transaminases and alkaline phosphatase less than or equal to 5 x the Upper Limit of Normal (ULN) obtained within 2 weeks prior to the first dose of study medication.
* The patient has adequate renal function as defined by serum creatinine less than or equal to 1.5 x ULN or calculated creatinine clearance (CrCl) >60 mL/minute, and urine dipstick for proteinuria <1+ (ie, either 0 or trace) obtained within 2 weeks prior to the first dose of study medication. If urine dipstick is greater than or equal to 1+, then a 24-hour urine for protein must demonstrate <500 mg of protein in 24 hours to allow participation in the study.
* The patient has adequate coagulation function as defined by International Normalized Ratio less than or equal to 1.5 and a Prothrombin time and partial thromboplastin time less than or equal to ULN obtained within 2 weeks prior to the first dose of study medication.
* The patient, if a woman of childbearing potential, agrees to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study. If a male and sexually active, the patient agrees to use effective contraception.

Exclusion Criteria:

* The patient has known Central Nervous System metastases. A head computed tomography (CT) is required within 4 weeks prior to the first dose of study medication (magnetic resonance imagines [MRIs] are also acceptable).
* The patient has received prior cetuximab therapy.
* The patient has received prior bevacizumab therapy.
* The patient has received prior systemic chemotherapy or radiation therapy at any time for lung cancer.
* Any concurrent malignancy other than basal cell skin cancer, or carcinoma in situ of the cervix. Patients with adequately treated cancers of other histologies who have been disease-free for more than 3 years prior to the first treatment dose are eligible.
* Concurrent treatment with other anti-cancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemoembolization, or targeted therapy.
* The patient has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The patient has a history of thrombotic or hemorrhagic disorders.
* The patient has uncontrolled hypertension (>150/100 mmHg) on a standard regimen of anti-hypertensive therapy.
* The patient is receiving chronic daily treatment with aspirin (>325 mg/day) or nonsteroidal anti-inflammatory agents known to inhibit platelet function.
* The patient is receiving treatment with dipyridamole (Persantine®), ticlopidine (Ticlid®), clopidogrel (Plavix®) and /or cilostazol (Pletal®).
* The patient is receiving anti-coagulation therapy. Prophylactic anti-coagulation of venous access devices is allowed. Caution should be taken on treating patients with low dose heparin or low molecular weight heparin for deep vein thrombosis (DVT) prophylaxis during treatment with bevacizumab as there may be an increased risk of bleeding.
* Patients with a history of gross hemoptysis (defined as bright red blood or greater than or equal to ½ teaspoon).
* The patient has a serious non-healing wound ulcer, bone fracture, or major surgical procedure within 30 days prior to first dose of study medication.
* Elective or planned major surgery to be performed during the course of the trial.
* The patient has a pre-existing neuropathy >grade 1.
* The patient, if a woman, is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (42):
- United States (42):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fountain Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grass Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfield, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evanston, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gurnee, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lambertville, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., High Point, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Langhorne, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willow Grove, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hilton Head Island, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mt. Pleasant, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnson City, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grapevine, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6): Cycles 1-6:
  * Cetuximab 400 mg/m² initial dose on day 1 and then 250 mg/m² given every week
  * Bevacizumab 15 mg/kg given on day 8 of every 3 week cycle
  * Paclitaxel 200mg/m² on day 1 of every 3 week cycle
  * Carboplatin AUC=6 min*mg/mL on day 1 of every 3 week cycle
  Patients who demonstrate a response or stable disease after six cycles of therapy may continue on weekly cetuximab monotherapy until disease progression, unacceptable toxicity, or another withdrawal criterion is met
Period: Overall Study
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3)
Started | 60 | 61
RECEIVED AT LEAST ONE DOSE OF STUDY DRUG | 58 | 58
Completed | 3 (Participants completed 6 cycles of treatment. Did not start subsequent weekly cetuximab monotherapy.) | 5 (Participants completed 6 cycles of treatment. Did not start subsequent weekly cetuximab monotherapy.)
Not Completed | 57 | 56
Not completed — Adverse Event | 13 | 13
Not completed — Death | 3 | 2
Not completed — Progressive disease | 33 | 34
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3) | Total
Number analyzed (Participants) | 60 | 61 | 121
Age Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.52) | 62.1 (8.97) | 62.8 (10.29)
Age, Customized [Number; unit: participants]
  < 65 years | 31 | 32 | 63
  ≥ 65 years | 29 | 29 | 58
Age, Customized [Number; unit: participants]
  < 70 years | 41 | 51 | 92
  ≥ 70 years | 19 | 10 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 35 | 34 | 69
Race/Ethnicity, Customized [Number; unit: participants]
  White | 53 | 53 | 106
  Black | 2 | 4 | 6
  Asian | 1 | 2 | 3
  Hispanic | 3 | 0 | 3
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 121
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Full Active | 24 | 29 | 53
    1 - Ambulatory, Restricted Strenuous Activity | 28 | 27 | 55
    Missing/Unknown | 8 | 5 | 13
Smoking Status [Number; unit: participants]
  Current | 17 | 11 | 28
  Past | 37 | 44 | 81
  Exposed to Second-hand Smoke | 2 | 1 | 3
  Not Exposed to Second-hand Smoke | 4 | 4 | 8
  Missing/Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization until the date of progression of disease (PD) or death from any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD ≥20% increase in sum of longest diameter of target lesions. Participants who are alive and without PD will be censored at the date of their last tumor assessment.
Time Frame: Randomization to PD or date of death from any cause up to 33.1 months
Population: Included all enrolled, randomized participants. All participants were analyzed as part of the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3)
Number analyzed (Participants) | 60 | 61
months | 6.05 [5.65 to 7.03] | 4.50 [4.01 to 5.42]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death. Participants who are alive will be censored on the last known alive date.
Time Frame: Randomization to the date of death from any cause up to 42.7 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3)
Number analyzed (Participants) | 60 | 61
months | 12.06 [9.40 to 19.25] | 11.63 [6.64 to 17.61]

3. Secondary Outcome: Percentage of Participants Achieving an Objective Overall Response (Overall Response Rate)
Description: The best objective overall response rate (ORR) is the percentage of randomized participants with a best overall response of complete response (CR) or partial response (PR), as classified by the investigator according to the RECIST guidelines. CR=disappearance of all target lesions; PR≥30% decrease in sum of longest diameter of target lesions. ORR is calculated as a total number of participants with CR or PR divided by the total number of participants treated in that arm, multiplied by 100. Participants with no post-baseline evaluation will be considered as a non-responder.
Time Frame: Randomization to measured progressive disease up to 31.8 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3)
Number analyzed (Participants) | 60 | 61
percentage of participants | 51.7 [39.0 to 64.3] | 44.3 [31.8 to 56.7]

4. Secondary Outcome: Duration of Overall Response
Description: The duration of response, in participants with best overall response of CR or PR, is measured from the date criteria are met for CR/PR (whichever is first recorded), until the first date that the criteria for PD is met or death. CR, PR, and PD, as classified by the investigator according to the RECIST guidelines. CR=disappearance of all target lesions; PR≥30% decrease in sum of longest diameter of target lesions; PD≥20% increase in sum of longest diameter of target lesions. Participants who are alive and without PD will be censored at the date of their last tumor assessment.
Time Frame: Time of first response to the first date of PD or death due to any cause up to 31.8 months
Population: Included all enrolled, randomized participants with a best overall response of CR or PR (responders). All participants were analyzed as part of the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3)
Number analyzed (Participants) | 31 | 27
months | 4.86 [4.30 to 7.16] | 3.94 [2.92 to 4.47]

5. Secondary Outcome: Percentage of Participants With Symptomatic Response (Symptom Response Rate)
Description: Functional Assessment of Cancer Therapy for Patients With Lung Cancer (FACT-L) measures domains of health-related quality of life (HR-QL): physical wellbeing (WB), social/family WB, emotional WB, functional WB, and additional lung cancer concerns. Symptom response (improvement) was defined as ≥2 point increase from baseline in the 7-item Lung cancer subscale (LCS) score maintained for 2 consecutive assessments. Scores range from 0-28 with higher scores indicating fewer symptoms. Patients with a score of >26 were not evaluable for symptom response, since a score of 28 is the maximum possible.
Time Frame: From date of partial response until progression of disease up to 31.8 months
Population: Included all enrolled, randomized participants with a score of ≤26 at baseline. All participants were analyzed as part of the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3)
Number analyzed (Participants) | 43 | 44
percentage of participants | 41.9 [27.1 to 56.6] | 38.6 [24.2 to 53.0]

ADVERSE EVENTS:
Description: Adverse events include all grades, regardless of severity or possible causality.
Arm/Group | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3)
Serious Adverse Events (participants affected / at risk) | 38/58 | 28/58
Other Adverse Events (participants affected / at risk) | 56/58 | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) (N=58) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3) (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (3)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Iga nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aortic embolus (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/6) (N=58) | Cetuximab + Bevacizumab + Paclitaxel + Carboplatin (6/3) (N=58)
Anaemia (Blood and lymphatic system disorders) | 21 (48) | 10 (12)
Neutropenia (Blood and lymphatic system disorders) | 17 (49) | 14 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (32) | 1 (3)
Palpitations (Cardiac disorders) | 3 (4) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 3 (4)
Vision blurred (Eye disorders) | 1 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (6)
Abdominal pain lower (Gastrointestinal disorders) | 4 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 22 (31) | 16 (20)
Diarrhoea (Gastrointestinal disorders) | 22 (29) | 14 (27)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 9 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 30 (53) | 23 (32)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 19 (37) | 23 (29)
Vomiting (Gastrointestinal disorders) | 12 (18) | 9 (11)
Asthenia (General disorders) | 7 (7) | 4 (6)
Catheter site pain (General disorders) | 0 (0) | 4 (4)
Chills (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 32 (61) | 28 (41)
Infusion related reaction (General disorders) | 1 (1) | 4 (13)
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 7 (10) | 4 (4)
Pain (General disorders) | 3 (4) | 4 (4)
Pyrexia (General disorders) | 7 (10) | 4 (5)
Hypersensitivity (Immune system disorders) | 2 (2) | 5 (6)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Fungal infection (Infections and infestations) | 3 (3) | 0 (0)
Localised infection (Infections and infestations) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 6 (9) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (15) | 6 (7)
Weight decreased (Investigations) | 10 (15) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 17 (23) | 18 (25)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 10 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 3 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 (40) | 13 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 16 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 11 (17)
Dizziness (Nervous system disorders) | 8 (13) | 5 (5)
Dysgeusia (Nervous system disorders) | 7 (9) | 7 (10)
Headache (Nervous system disorders) | 8 (8) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 17 (31) | 12 (16)
Paraesthesia (Nervous system disorders) | 2 (2) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (12) | 8 (12)
Tremor (Nervous system disorders) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (5) | 10 (10)
Confusional state (Psychiatric disorders) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 10 (11) | 9 (9)
Insomnia (Psychiatric disorders) | 11 (11) | 13 (15)
Dysuria (Renal and urinary disorders) | 3 (3) | 3 (3)
Proteinuria (Renal and urinary disorders) | 8 (9) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 13 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 8 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (26) | 22 (27)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 45 (96) | 40 (74)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (20) | 10 (11)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (15)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (4)
Skin fissures (Skin and subcutaneous tissue disorders) | 3 (6) | 3 (6)
Flushing (Vascular disorders) | 4 (5) | 1 (2)
Hypertension (Vascular disorders) | 3 (4) | 10 (11)
Hypotension (Vascular disorders) | 7 (8) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days